CLINICAL TRIAL: NCT04262570
Title: Evaluation of Therapeutic Response in Spinal Muscular Atrophy Using Multispectral Optoacoustic Tomography (MSOT) and Magnetic Resonance Imaging (MRI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 453_19B
Record Dates: First submitted 2020-01-27; First posted 2020-02-10 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Muscular Diseases; Spinal Muscular Atrophy
Keywords: Muscular Diseases; Spinal Muscular Atrophy (SMA); Multispectral Optoacoustic Tomography (MSOT); Magnetic Resonance Imaging (MRI)
MeSH Terms: conditions — Muscular Diseases; Muscular Atrophy, Spinal | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMA patients (therapy arm) (Experimental): * Multispectral Optoacoustic Tomography (MSOT) of muscles (left and right, total 4 sites) leg proximal: Musculus quadriceps, distal: Musculus triceps surae arm proximal: Musculus biceps, distal: forearm flexors;
  * Magnetic Resonance Imaging (MRI) of lower leg
  * Physical assessment/milestones: expanded Hammersmith functional motor scale (HFMSE)/ Revised Upper Limb Module (RULM)/ 6-minute-walking-test (6-MWT)
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT) and Magnetic Resonance Imaging (MRI)
- SMA patients (control arm) (Active Comparator): * Multispectral Optoacoustic Tomography (MSOT) of muscles (left and right, total 4 sites) leg proximal: Musculus quadriceps, distal: Musculus triceps surae arm proximal: Musculus biceps, distal: forearm flexors;
  * Magnetic Resonance Imaging (MRI) of lower leg
  * Physical assessment/milestones: expanded Hammersmith functional motor scale (HFMSE)/ Revised Upper Limb Module (RULM)/ 6-minute-walking-test (6-MWT)
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT) and Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Device: Multispectral Optoacoustic Tomography (MSOT) and Magnetic Resonance Imaging (MRI) — Non-invasive transcutaneous imaging of molecular muscle components

SUMMARY:
This study aims to refine the capability of Multispectral Optoacoustic Tomography (MSOT) and Magnet Resonance Imaging (MRI) to characterise the molecular composition of muscle tissue non-invasively and to evaluate the therapeutic response in patients with spinal muscular atrophy (SMA) over time.

DETAILED DESCRIPTION:
SMA is an autosomal-recessive disorder, characterized by progressive muscle weakness and atrophy with an incidence of 1/10,000. The condition is caused by a homozygous deletion or mutation in the survival motor neuron 1 (SMN1), resulting in reduced expression of the survival motor neuron (SMN) protein. This leads to the degeneration of motor neurons in the spinal cord and brain stem. A nearby related gene, survival motor neuron 2 (SMN2), could partially compensate the loss of SMN1. Individuals with a higher copy number of SMN2 do in general have a milder phenotype. New therapeutic approaches, e.g. nusinersen (spinraza©), an antisense oligonucleotide medication that modulates pre-messenger RNA splicing of the survival motor neuron 2 (SMN2) gene, are promising to help the formerly incurable disease. However, most clinical trials lack primary outcomes other than clinical testing. Preliminary work shows that new methods such as multispectral optoacoustic tomography (MSOT) and magnetic resonance imaging (MRI) detect tissue changes very sensitively. Multispectral optoacoustic tomography (MSOT) is capable of visualizing the distribution of endogenous absorbers by initiating laser-induced thermoelastic expansion and detection of resulting pressure waves. This imaging technique enables the label-free detection and quantification of different endogenous chromophores. In addition to this technology, MRI imaging has advanced in the field of muscle diseases, with 23Na-MRI being the first example. With both methods, the molecular composition of muscle tissue can be determined non-invasively and quantitatively at the same time. In this first pilot study on patients with SMA, the investigators will now assess whether the differences in the muscle composition of SMA patients with or without therapy can be quantified and whether they can be used simultaneously as markers during therapy with nusinersen (spinraza©) . Ideally, both techniques can complement or validate each other. In the future, this could generate a completely new, non-invasive method for evaluating endogenous biomarkers for therapy response.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed SMA type III
* From age 14
* Willingness and ability to participate, sufficient knowledge of the german language to understand the declaration of consent, or if not possible, information of the patient in his/her mother tongue or English
* High probability that the patients will be able to fully participate in the study (defined by the ability to lie still for about 1 hour and follow any breathing commands) For therapy arm: • Medical indication for Spinraza® therapy; start of study before first administration Spinraza® administration For control arm: • No medical indication for Spinraza® therapy

Exclusion Criteria:

* Pregnancy
* Tattoo on the skin area to be examined
* General contraindications for MRT examinations
* Electrical implants like pacemakers or perfusion pumps
* Pronounced claustrophobia
* Study participants with ferromagnetic or electrically conductive implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, heart valves with metal parts, metal splinters, tattoos next to the eye, symmetrical tattoos on the extremities or steel implants must consult the study physician; they may not be able to be examined (relative contraindications for MRI).
* Non-approved concomitant medication: strongly sedating medication must be excluded, as intensive monitoring of bodily functions during ongoing imaging cannot be guaranteed and the active participation of the test person might be necessary.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of muscle structure under therapy and change from baseline over time | 3 time points (at 0,2, and 12 months)
  Comparison of the molecular muscle structure determined by MSOT and MRI in patients with SMA with and without treatment and evaluation of changes from baseline over time

SECONDARY OUTCOMES:
Muscular lipid content | 3 time points (at 0,2, and 12 months)
  Quantitative lipid signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with SMA with and without therapy and change over time Units: arbitrary units (a.u.)
Muscular collagen content | 3 time points (at 0,2, and 12 months)
  Quantitative collagen signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with SMA with and without therapy and change over time Units: arbitrary units (a.u.)
Muscular hemo-/myoglobin content | 3 time points (at 0,2, and 12 months)
  Quantitative hemo/myoglobin signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with SMA with and without therapy and change over time Units: arbitrary units (a.u.)
Muscular de-/oxygenated hemo-/myoglobin content | 3 time points (at 0,2, and 12 months)
  Quantitative de-/oxygenated hemo-/myoglobin signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with SMA with and without therapy and change over time Units: arbitrary units (a.u.)
Ratio of lipid to hemo/myoglobin signal or collagen to hemo/myoglobin signal | 3 time points (at 0,2, and 12 months)
  Ratio of quantitative lipid signal to hemo/myoglobin signal or collagen signal to hemo/myoglobin signal derived by transcutaneous Multispectral Optoacoustic Tomography (MSOT) in patients with SMA with and without therapy and change over time
T1 relaxation time | 3 time points (at 0,2, and 12 months)
  T1 relaxation time determined by Magnetic Resonance Imaging (MRI) in patients with SMA with and without therapy and change over time
T2 relaxation time | 3 time points (at 0,2, and 12 months)
  T2 relaxation time determined by Magnetic Resonance Imaging (MRI) in patients with SMA with and without therapy and change over time
Fat-water percentage | 3 time points (at 0,2, and 12 months)
  Fat-water percentage determined by Magnetic Resonance Imaging (MRI) in patients with SMA with and without therapy and change over time
Sodium concentration | 3 time points (at 0,2, and 12 months)
  Sodium concentration determined by Magnetic Resonance Imaging (MRI) in patients with SMA with and without therapy and change over time
Correlation of MSOT data with therapy status | 3 time points (at 0,2, and 12 months)
  Correlation of the quantitative lipid/collagen/hemo/myoglobin and de-/oxygenated hemo-/myoglobin content determined by MSOT in patients with and without therapy and evaluation of change over time
Correlation of MSOT data with clinical data (age/disease duration) | 3 time points (at 0,2, and 12 months)
  Correlation of lipid/collagen/haemo/myoglobin and de-/oxygenated hemo-/myoglobin content determined by MSOT with disease duration/patient age and evaluation of change over time
Correlation of MSOT data with physical assessment (HFMSE/RULM/6-MWT) | 3 time points (at 0,2, and 12 months)
  Correlation of lipid/collagen/haemo/myoglobin and de-/oxygenated hemo-/myoglobin content determined by MSOT with HFMSE/Revised Upper Limb Module/6-MWT and evaluation of change over time
Correlation of MRI data with therapy status | 3 time points (at 0,2, and 12 months)
  Correlation of T1 relaxation time/T2 relaxation time/fat water portion/sodium concentration in patients with and without therapy and evaluation of change over time
Correlation of MRI data with clinical data (age/disease duration) | 3 time points (at 0,2, and 12 months)
  Correlation of T1 relaxation time/T2 relaxation time/fat water portion/sodium concentration with disease duration and patient age and evaluation of change over time
Correlation of MRI data with physical assessment (HFMSE/RULM/6-MWT) | 3 time points (at 0,2, and 12 months)
  Correlation of T1 relaxation time/T2 relaxation time/fat water portion/sodium concentration with HFMSE/Revised Upper Limb Module/6-MWT and evaluation of change over time
Correlation of MSOT data and MRI data | 3 time points (at 0,2, and 12 months)
  Correlation of MSOT determined lipid/collagen/haemo/myoglobin and de-/oxygenated hemo-/myoglobin content and MRI derived T1 relaxation time/T2 relaxation time/fat water portion/sodium concentration and evaluation of change over time
Side differences | 3 time points (at 0,2, and 12 months)
  Measurement of the signal differences in right / left comparison derived by Multispectral Optoacoustic Tomography (MSOT) and Magnetic Resonance Imaging (MRI) and evaluation of change over time

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinand Knieling, MD, Principal Investigator — University Hospital Erlangen, Department of Pediatric and Adolescent Medicine; Matthias Türk, MD, Principal Investigator — University Hospital Erlangen, Department of Neurology; Armin Nagel, MD, Principal Investigator — University Hospital Erlangen, Department of Radiology
Locations (1):
- University Hospital Erlangen, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary publication, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request as follows:
  * Individual participant data will not be available
  * Study Protocol and Statistical Analysis Plan will be available
  * The data will be available beginning 9 months and ending 36 months following article publication.
  * The data will be available to researchers who provide a methodologically sound proposal.
  * The data will be available for individual participant data meta-analysis, only.
  * Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at https://www.uk-erlangen.de.
  Restrictions may apply due to patient privacy and the General Data Protection Regulation.

DOCUMENTS (1):
  • Study Protocol (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT04262570/Prot_001.pdf